CLINICAL TRIAL: NCT04477174
Title: Validity and Reliability of the Turkish Translation of the Yale Pharyngeal Residue Severity Rating Scale (YPRSRS-T)
Brief Title: Validity and Reliability of the Turkish Translation of the Yale Pharyngeal Residue Severity Rating Scale
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Yavuz Atar, Associate Professor, M.D., Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 308
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Swallowing Disorder; Validation; Pharyngeal Dysphagia
Keywords: Pharyngeal; residue; swallow; scale; Yale
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Twelve health professionals randomised assign to as equally count. The participants match between the images with scale scores. After 2 weeks, the participants match again.
- Group B: Twelve health professionals randomised assign to as equally count. The participants match between the images with scale scores.

SUMMARY:
Purpose of the study is the validity and reliability of the Turkish version of the Yale Pharyngeal Residue Severity Rating Scale (YPRSRS-T), so that it would be used as an assessment tool for dysphagia patients.

DETAILED DESCRIPTION:
The swallow function is a multidirectional process that depends on complex neuro-muscular network. The function can be evaluated using instrumental, such as fibreoptic endoscopic evaluation of swallowing (FEES), videofluoroscopy, or well structured scales. There are many questionnaire and scales for assessment of swallow but very few have been validated. The study will assess the construct validity and reliability of the Turkish version of Pharyngeal Residue Severity Rating Scale as known as Yale Pharyngeal Residue Severity Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* at least having undergraduate education on health profession
* agree to participant

Exclusion Criteria:

* out of age 18-70 years
* out of having undergraduate education
* mental disorder
* cognitive limitations
* visual limitations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health professionals
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Validation of Pharyngeal Residue Severity Rating Scale | 2 months
  To match between Fiberoptic Endoscopic Evaluation of Swallowing Images with Yale Pharyngeal Residue Severity Rating Scale Scores by health professionals. High match scores give high reliability, low match scores give low reliability. Match scores were compared and evaluated as statistically. High match score is better, low score is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Melis Ece Arkan Ararat, MD, Principal Investigator — University of Health Sciences, Prof Dr Cemil Tascioglu City Hospital; Ugur Uygan, MD, Principal Investigator — University of Health Sciences, Prof Dr Cemil Tascioglu City Hospital
Locations (1):
- Prof Dr Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No